CLINICAL TRIAL: NCT02606422
Title: Effects of Transcranial Direct Current Stimulation (tDCS) in Spoken and Written Production in Primary Progressive Aphasia (PPA)
Brief Title: tDCS Intervention in Primary Progressive Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA_00071337; R01DC014475 (NIH)
Record Dates: First submitted 2015-11-11; First posted 2015-11-17 (Estimated); Results first posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Primary Progressive Aphasia; MCI; FTD
Keywords: transcranial direct current stimulation (tDCS); neurodegeneration; language therapy; Primary Progressive Aphasia (PPA)
MeSH Terms: conditions — Aphasia, Primary Progressive; Nerve Degeneration | interventions — Speech Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active HD-tDCS plus Speech-Language Therapy (Experimental): Active HD-tDCS will be applied at the beginning of 45min speech-language therapy session and will last for 20 min.
  Interventions: Device: Active HD-tDCS plus Speech-Language Therapy
- Sham plus Speech-Language Therapy (Sham Comparator): Sham HD-tDCS will be applied at the beginning of 45min speech-language therapy session.
  Interventions: Device: Sham plus Speech-Language Therapy

INTERVENTIONS:
Device: Active HD-tDCS plus Speech-Language Therapy — Stimulation will be delivered by a battery-driven constant current stimulator. The electrical current will be administered to a pre-specified region of the brain (inferior frontal gyrus). The stimulation will be delivered at an intensity of 2mA (estimated current density 0.04 mA/cm2; estimated total charge 0.048C/cm2) in a ramp-like fashion for a maximum of 20 minutes. Speech-language therapy will be oral and written naming.
  Arms: Active HD-tDCS plus Speech-Language Therapy
Device: Sham plus Speech-Language Therapy — Speech-language therapy will be administered during sham stimulation. Current will be administered in a ramp-line fashion but after the ramping the intensity will drop to 0 mA. Speech-language therapy will be oral and written naming.
  Arms: Sham plus Speech-Language Therapy

SUMMARY:
Primary progressive aphasia (PPA) is a neurodegenerative disease that affects first and foremost language abilities. Mild cognitive impairment (MCI) is slowly progressive decline in a single domain of cognition (e.g. language) not attributable to motor or sensory loss, without impediment of social or occupational function. MCI can be an early sign of neurodegenerative disease, or can be due to normal aging. When language is the prominent affected domain in MCI, the person may later meet criteria for PPA or may progress to the clinical syndrome of Alzheimer's dementia. Spelling, naming, and working memory (e.g. repetition) are among the language abilities affected early in the course of PPA or language-centered MCI, and different variants have distinct deficits in these domains. This research project investigates the behavioral and neuromodulatory effects of high definition transcranial direct current stimulation (HD-tDCS) during language therapy in PPA participants over time. Anodal HD-tDCS targeting the left inferior frontal gyrus (IFG) administered in combination with language therapy is expected to be more beneficial when compared to language therapy alone. It will 1) improve language performance or decrease rate of decline, 2) have better-sustained effects at 2 weeks and 2 months post-treatment, and 3) produce generalization to untrained language items and some other cognitive functions. Resting-state fMRI, diffusion tensor imaging (DTI), and volumetric data are also collected to investigate changes in functional brain connectivity associated with HD-tDCS in individuals with PPA. A better understanding of the therapeutic and neuromodulatory mechanisms of HD-tDCS as an adjunct to language therapy in PPA may have a significant impact on the development of effective therapies for PPA and MCI, and may offer insight into ways of impeding neurodegeneration that may improve patients' quality of life, as well as extend their ability to work and manage their affairs.

DETAILED DESCRIPTION:
A. Evaluation Tasks

Language Tasks:

Participants will be administered baseline language and cognitive tasks, including 1 or more of the following, depending on their residual language and cognitive skills:

a) writing to dictation b) oral spelling c) oral and written naming of pictures d) word-picture matching f) written and oral picture description g) digit span h) spatial span i) verbal learning j) grammatical sentence production k) oral word repetition l) sentence comprehension

Quality of Life questionnaires:

Participants will be administered standardized and non-standardized quality-of-life questionnaires before, after, and at follow-up intervals of each experimental period. The purpose of these questionnaires is to assess whether the proposed interventions have affected participants' well-being and the general quality of their life.

B. Spoken and Written Word Production Therapy Interventions

Individuals with PPA will receive spoken and written word production intervention tailored to their degree of deficit. Two interventions (basic and advanced) will be implemented, treating the main lexical retrieval deficits in PPA, in oral and written modalities. The goal of the combined interventions is to promote interaction between phonological and orthographic representations and processes in the remediation of lexical retrieval deficits that are prominent in all PPA subtypes.

C. Assessment of Language Therapy Tasks:

Follow-up assessment will probe all sets of trained phoneme-grapheme correspondences, words, or other stimuli (e.g. sentences) to identify whether or not the patient has retained knowledge of the trained items. Differences in baseline measures in pre- and post-therapy accuracy for phoneme-grapheme correspondences for each patient will be evaluated using the following: percentages of total number of points correct, arithmetic differences between percentage scores, and permutation tests (Pearson's chi-square test; Fisher's exact test).

C. HD-tDCS Methods:

Participants will take part in 10-15 consecutive training sessions (3-5 per week), separated by 2 months. Anodal HD-tDCS has typically been shown to up-regulate neuronal excitability and produce enhancement of behavioral performance. A Soterix-CT device will be delivering current at an intensity of 1-2 milliamps(mA) (estimated current density 0.04 mA/cm2; estimated total charge 0.048C/cm2) for a maximum of 20 minutes in the HD-tDCS groups and for a maximum of 30 seconds in the Sham group. For both interventions (HD-tDCS and Sham) the electrical current will be increased in a ramp-like fashion at the onset of the stimulation eliciting a transient tingling sensation on the scalp that usually disappears over seconds.

D. Imaging Methods:

Imaging will be performed at the beginning of enrollment, before and after each 12-to-15-day HD-tDCS treatment, and at follow-up intervals for up to 8 time points per individual on a 3T Philips system, and will consist of resting-state fMRI (rsfMRI), MPRAGE, and diffusion tensor imaging (DTI). Each scanning session will last approximately 1 hour.

E. Statistical Analyses:

In the within-subject crossover protocol, each participant will be administered three experimental conditions: Control (natural progression), IFG HD-tDCS+language (henceforth abbr. HD-tDCS treatment (word production) and sham HD-tDCS+language (henceforth abbr. sham treatment). To achieve an accurate estimate of degeneration and rate of decline in each participant at their particular stage of the disease progression, each participant will first be enrolled in the control condition (natural progression), such that for the first 12 weeks they will not receive any therapy. Then the participant will receive either the HD-tDCS treatment followed by sham, or vice versa. All analyses, behavioral and imaging, will be under the oversight of the study statisticians.

F. Study duration and number of study visits required of research participants.

Before any intervention, participants will be enrolled in a control condition for 12 weeks during which no therapy will be provided to enable us to assess their personal decline rate. After this period they will be randomly assigned to either sham or HD-tDCS experimental conditions. After 1-3 weeks of HD-tDCS application (3-5 sessions in a week, 10-15 sessions per stimulation site) there will be an interval of approximately 2 months and then we will implement the other two HD-tDCS conditions in a within-subject cross-over design. Participants will be followed up at 2-week and 2-month follow-up intervals.

G. Blinding, including justification for blinding or not blinding the trial, if applicable.

Participants will be blinded to the application of anodal or sham HD-tDCS. To achieve blinding, all participants will be fitted with the HD-tDCS electrodes placed over the left inferior frontal gyrus. The Soterix-CT device will be used for double-blinding purposes.

H. Justification of why participants will not receive routine care or will have current therapy stopped

Participation in this study will not disrupt any current care or therapy.

I. Justification for inclusion of a placebo or non-treatment group

All participants will undergo active and sham conditions, thus serving as their own control.

J. Definition of treatment failure or participant removal criteria

Participants will be removed from the study if they are unable to comply with task instructions or tolerate the HD-tDCS procedure.

K. Description of what happens to participants receiving therapy when the study ends or if a participant's participation in the study ends prematurely

When the study ends participants will continue to receive management with their neurologist as usual. If a patient's participation in the study ends prematurely s/he will still receive care as before. In sum, termination of the study or termination of participation in it will not affect the regular therapy he or she may be receiving.

L. Qualification of investigators:

The PI and co-investigators have extensive research and clinical experience with all study tasks: behavioral language therapy (including spelling, naming, and repetition therapy. The investigators have already published a tDCS study on the behavioral results for the improvement of spelling abilities.

ELIGIBILITY:
Inclusion Criteria:

* Must be clinically diagnosed with semantic variant PPA (svPPA), non-fluent variant PPA (nfvPPA), or logopenic variant PPA (lvPPA), unclassifiable PPA, or MCI. Diagnosis will be based on neuropsychological testing, language testing (most commonly the Western Aphasia Battery), MRI and clinical assessment.
* Must be right-handed.
* Must be speakers of English.
* Must have at least 9th grade education.

Exclusion Criteria:

* Uncorrected visual or hearing impairment by self report.
* Stroke/other premorbid neurological disorder affecting the brain.
* Any other language-based learning disorder other than PPA.
* Inability to follow directions for baseline tasks.
* Western Aphasia Battery Aphasia Quotient (AQ) <30 (indicating severe language impairment).

Exclusion Criteria for MRI Participation:

* Severe claustrophobia.
* Cardiac pacemakers or ferromagnetic implants.
* Pregnant women.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-04; Primary Completion 2023-07-12 (Actual); Study Completion 2023-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyrana Tsapkini, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Tsapkini K, Frangakis C, Gomez Y, Davis C, Hillis AE. Augmentation of spelling therapy with transcranial direct current stimulation in primary progressive aphasia: Preliminary results and challenges. Aphasiology. 2014;28(8-9):1112-1130. doi: 10.1080/02687038.2014.930410. PMID 26097278
- [Background] Tippett DC, Hillis AE, Tsapkini K. Treatment of Primary Progressive Aphasia. Curr Treat Options Neurol. 2015 Aug;17(8):362. doi: 10.1007/s11940-015-0362-5. PMID 26062526
- [Result] Tsapkini K, Webster KT, Ficek BN, Desmond JE, Onyike CU, Rapp B, Frangakis CE, Hillis AE. Electrical brain stimulation in different variants of primary progressive aphasia: A randomized clinical trial. Alzheimers Dement (N Y). 2018 Sep 5;4:461-472. doi: 10.1016/j.trci.2018.08.002. eCollection 2018. PMID 30258975
- [Derived] Wang Z, Ficek BN, Webster KT, Herrmann O, Frangakis CE, Desmond JE, Onyike CU, Caffo B, Hillis AE, Tsapkini K. Specificity in Generalization Effects of Transcranial Direct Current Stimulation Over the Left Inferior Frontal Gyrus in Primary Progressive Aphasia. Neuromodulation. 2023 Jun;26(4):850-860. doi: 10.1016/j.neurom.2022.09.004. Epub 2022 Oct 28. PMID 37287321
- [Derived] Herrmann O, Ficek B, Webster KT, Frangakis C, Spira AP, Tsapkini K. Sleep as a predictor of tDCS and language therapy outcomes. Sleep. 2022 Mar 14;45(3):zsab275. doi: 10.1093/sleep/zsab275. PMID 34875098
- [Derived] Tao Y, Ficek B, Rapp B, Tsapkini K. Different patterns of functional network reorganization across the variants of primary progressive aphasia: a graph-theoretic analysis. Neurobiol Aging. 2020 Dec;96:184-196. doi: 10.1016/j.neurobiolaging.2020.09.007. Epub 2020 Sep 8. PMID 33031971
- See also: Tsapkini 2014 — http://www.ncbi.nlm.nih.gov/pubmed/26097278
- See also: Tsapkini 2015 — http://www.ncbi.nlm.nih.gov/pubmed/26062526

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 61 patients were consented for eligibility between the study start date and end date at our lab located at Johns Hopkins Hospital.
Pre-assignment Details: All 61 participants that were consented started a 12-week natural progression observation where they did not recieve any therapy. After the 12-week period, 37 participants were randomized. Of those not randomized,13 had a primary deficit of apraxia of speech, 7 chose not to participate, 1 did not have measureable language deficits, 3 chose to participate in another trial.
Groups:
- Active HD-tDCS Plus Speech-Language Therapy, Then Sham Plus Speech-Language Therapy: Participants first received active tDCS with speech therapy for two weeks. Active high-Definition transcranial Direct Current Stimulation (HD-tDCS) was applied at the beginning of 45 min speech-language therapy session and lasted for 20 min. The electrical current was administered to a pre-specified region of the brain (inferior frontal gyrus). The stimulation was delivered at an intensity of 2 miliamps (mA) (estimated current density 0.04 mA/cm2; estimated total charge 0.048 coulombs (C)/cm2) in a ramp-like fashion for a maximum of 20 minutes. Speech-language therapy consisted of oral and written naming. After a washout period of 3 months, they then received sham tDCS plus speech therapy for 2 weeks. Speech-language therapy will be administered during sham stimulation. Current was administered in a ramp-line fashion but after the ramping, the intensity dropped to 0 mA
- Sham Plus Speech-Language Therapy, Then Active HD-tDCS Plus Speech-Language Therapy: Participants first received sham tDCS with speech therapy for 2 weeks. Sham HD-tDCS was applied at the beginning of 45 min speech-language therapy session and lasted for 20 min. The electrical current was administered to a pre-specified region of the brain (inferior frontal gyrus). Speech-language therapy will be administered during sham stimulation. Current was administered in a ramp-line fashion but after the ramping the intensity dropped to 0 mA. After a washout period of 3 months, they then received active tDCS plus speech therapy for two weeks. The stimulation was delivered at an intensity of 2mA (estimated current density 0.04 mA/cm2; estimated total charge 0.048C/cm2) in a ramp-like fashion for a maximum of 20 minutes. Speech-language therapy consisted of oral and written naming.
Period: Intervention Phase 1 (3 Weeks)
Arm/Group | Active HD-tDCS Plus Speech-Language Therapy, Then Sham Plus Speech-Language Therapy | Sham Plus Speech-Language Therapy, Then Active HD-tDCS Plus Speech-Language Therapy
Started | 20 | 17
Completed | 20 | 17
Not Completed | 0 | 0
Period: Phase 1: Immediate Follow up
Arm/Group | Active HD-tDCS Plus Speech-Language Therapy, Then Sham Plus Speech-Language Therapy | Sham Plus Speech-Language Therapy, Then Active HD-tDCS Plus Speech-Language Therapy
Started | 20 (Two participants dropped out) | 17
Completed | 18 | 17
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: Phase 1, 2-Week Follow-up (Washout)
Arm/Group | Active HD-tDCS Plus Speech-Language Therapy, Then Sham Plus Speech-Language Therapy | Sham Plus Speech-Language Therapy, Then Active HD-tDCS Plus Speech-Language Therapy
Started | 18 | 17
Completed | 16 | 17
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: Phase 1 2-Month Follow-up (Washout)
Arm/Group | Active HD-tDCS Plus Speech-Language Therapy, Then Sham Plus Speech-Language Therapy | Sham Plus Speech-Language Therapy, Then Active HD-tDCS Plus Speech-Language Therapy
Started | 16 | 17
Completed | 15 | 16
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Intervention Phase 2 (3 Weeks)
Arm/Group | Active HD-tDCS Plus Speech-Language Therapy, Then Sham Plus Speech-Language Therapy | Sham Plus Speech-Language Therapy, Then Active HD-tDCS Plus Speech-Language Therapy
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0
Period: Phase 2: Immediate Follow-up
Arm/Group | Active HD-tDCS Plus Speech-Language Therapy, Then Sham Plus Speech-Language Therapy | Sham Plus Speech-Language Therapy, Then Active HD-tDCS Plus Speech-Language Therapy
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0
Period: Phase 2, 2-Week Follow-up (Washout)
Arm/Group | Active HD-tDCS Plus Speech-Language Therapy, Then Sham Plus Speech-Language Therapy | Sham Plus Speech-Language Therapy, Then Active HD-tDCS Plus Speech-Language Therapy
Started | 15 | 16 (One participant dropped out)
Completed | 15 | 15
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Phase 2: 2-Month Follow-up (Washout)
Arm/Group | Active HD-tDCS Plus Speech-Language Therapy, Then Sham Plus Speech-Language Therapy | Sham Plus Speech-Language Therapy, Then Active HD-tDCS Plus Speech-Language Therapy
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active HD-tDCS Plus Speech-Language Therapy, Then Sham Plus Speech-Language Therapy: Participants first received active tDCS with speech therapy for two weeks. Active HD-tDCS was applied at the beginning of 45 min speech-language therapy session and lasted for 20 min. The electrical current was administered to a pre-specified region of the brain (inferior frontal gyrus). The stimulation was delivered at an intensity of 2mA (estimated current density 0.04 mA/cm2; estimated total charge 0.048C/cm2) in a ramp-like fashion for a maximum of 20 minutes. Speech-language therapy consisted of oral and written naming. After a washout period of 3 months, they then received sham tDCS plus speech therapy for 2 weeks. Speech-language therapy will be administered during sham stimulation. Current was administered in a ramp-line fashion but after the ramping, the intensity dropped to 0 mA
- Total: Total of all reporting groups
Arm/Group | Active HD-tDCS Plus Speech-Language Therapy, Then Sham Plus Speech-Language Therapy | Sham Plus Speech-Language Therapy, Then Active HD-tDCS Plus Speech-Language Therapy | Total
Number analyzed (Participants) | 20 | 17 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.45 (7.40) | 68.82 (7.05) | 67.45 (7.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 11 | 9 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 17 | 37

OUTCOME MEASURES:

1. Primary Outcome: Absolute Percent Change in Written Naming (Trained Items)
Description: The primary outcome measure was the absolute percentage change in the number of correct letters in the written response, compared to the target response in the trained word lists. This calculation reflects the change in accuracy between two timepoints.
  For letter accuracy scoring, a rule-based system was used where each letter was assigned one point if correct. Points were deducted for errors such as deletions, additions, substitutions, transpositions, or movements of letters. A second reviewer independently scored the responses and resolved any discrepancies through discussion to ensure consensus. Interrater reliability for letter accuracy scoring was 95%.
  Average letter accuracy per word was calculated for all trained items. Then the absolute percentage change was calculated by subtracting the earlier time point value (e.g., baseline) from the later one (e.g., immediately after treatment, 2 weeks post, and 2 months post), reflecting the change in accuracy.
Time Frame: Change from Baseline to Immediately after treatment (3 weeks), 2 weeks post treatment (5 weeks), and 2 months post-treatment (11 weeks) for each period of intervention
Population: Participants who completed Written Naming
Measure: Mean (Standard Error); unit: absolute percent change
Groups:
- Active tDCS Plus Speech-Language Therapy: Active tDCS will be applied at the beginning of 45min speech-language therapy session and will last for 20 min.
  Active tDCS plus Speech-Language Therapy: Stimulation will be delivered by a battery-driven constant current stimulator. The electrical current will be administered to a pre-specified region of the brain (inferior frontal gyrus). The stimulation will be delivered at an intensity of 2mA (estimated current density 0.04 mA/cm2; estimated total charge 0.048C/cm2) in a ramp-like fashion for a maximum of 20 minutes. Speech-language therapy will be oral and written naming.
Arm/Group | Active tDCS Plus Speech-Language Therapy | Sham Plus Speech-Language Therapy
Number analyzed (Participants) | 34 | 31
absolute percent change
  Phase 1: Change from baseline to immediately after treatment: number analyzed (Participants) | 19 | 16
  Phase 1: Change from baseline to immediately after treatment | 39.4 (5.1) | 28.4 (5.2)
  Phase 1: change from baseline to 2-weeks post treatment: number analyzed (Participants) | 18 | 16
  Phase 1: change from baseline to 2-weeks post treatment | 33.1 (4.7) | 20.0 (5.1)
  Phase 1: change from baseline to 2-months post treatment. (Baseline for Phase 2): number analyzed (Participants) | 16 | 16
  Phase 1: change from baseline to 2-months post treatment. (Baseline for Phase 2) | 27.5 (5.5) | 11.7 (2.7)
  Phase 2: Change from baseline to immediate follow-up: number analyzed (Participants) | 15 | 15
  Phase 2: Change from baseline to immediate follow-up | 27.0 (5.4) | 25.5 (6.2)
  Phase 2:change from baseline to 2-weeks post treatment: number analyzed (Participants) | 14 | 14
  Phase 2:change from baseline to 2-weeks post treatment | 13.2 (4.9) | 13.2 (6.7)
  Phase 2: change from baseline to 2-months post treatment: number analyzed (Participants) | 14 | 15
  Phase 2: change from baseline to 2-months post treatment | 9.1 (4.1) | 8.9 (4.6)

2. Primary Outcome: Absolute Percent Change in Written Naming (Untrained Items)
Description: The primary outcome measure was the absolute percentage change in the number of correct letters in the written response, compared to the target response in the untrained word lists.This calculation reflects the change in accuracy between two timepoints.
  For letter accuracy scoring, a rule-based system was used where each letter was assigned one point if correct. Points were deducted for errors such as deletions, additions, substitutions, transpositions, or movements of letters. A second reviewer independently scored the responses and resolved any discrepancies through discussion to ensure consensus. Interrater reliability for letter accuracy scoring was 95%.
  Average letter accuracy per word was calculated for all untrained items. Then the absolute percentage change was calculated by subtracting the earlier time point value (e.g., baseline) from the later one (e.g., immediately after treatment, 2 weeks post, and 2 months post), reflecting the change in accuracy.
Time Frame: as for outcome 1
Population: Participants who completed written naming
Measure: Mean (Standard Error); unit: absolute percent change
Groups:
- Sham tDCS Plus Speech-Language Therapy: Sham HD-tDCS will be applied at the beginning of 45min speech-language therapy session.
  Sham plus Speech-Language Therapy: Speech-language therapy will be administered during sham stimulation. Current will be administered in a ramp-line fashion but after the ramping the intensity will drop to 0 mA. Speech-language therapy will be oral and written naming.
Arm/Group | Active tDCS Plus Speech-Language Therapy | Sham tDCS Plus Speech-Language Therapy
Number analyzed (Participants) | 34 | 31
absolute percent change
  Phase 1: change from baseline immediately after treatment: number analyzed (Participants) | 19 | 16
  Phase 1: change from baseline immediately after treatment | 14.6 (2.7) | 9.6 (2.3)
  Phase 1: change from baseline 2-weeks post treatment: number analyzed (Participants) | 18 | 16
  Phase 1: change from baseline 2-weeks post treatment | 15.6 (3.9) | 6.6 (3.4)
  Phase 1: change from baseline 2-months post treatment. (Baseline for Phase 2): number analyzed (Participants) | 16 | 16
  Phase 1: change from baseline 2-months post treatment. (Baseline for Phase 2) | 17.3 (3.6) | 3.0 (3.0)
  Phase 2: change from baseline immediately after treatment: number analyzed (Participants) | 15 | 15
  Phase 2: change from baseline immediately after treatment | 9.9 (2.6) | 5.4 (2.5)
  Phase 2: change from baseline 2-weeks post treatment: number analyzed (Participants) | 14 | 14
  Phase 2: change from baseline 2-weeks post treatment | 7.3 (3.9) | 0.7 (2.2)
  Phase 2: change from baseline 2-months post treatment: number analyzed (Participants) | 14 | 15
  Phase 2: change from baseline 2-months post treatment | 9.9 (1.9) | -3.4 (2.7)

3. Primary Outcome: Absolute Percent Change in Oral Naming (Trained Items)
Description: The percent accuracy for each participant's trained oral naming list was calculated, with scores ranging from 0% to 100%. A score of 0% indicates no correct responses, while 100% represents perfect accuracy. Higher percentages reflect better performance. To assess changes in performance from pre- to post-treatment, the percent accuracy for untrained items was compared before and after the intervention. The absolute percentage change was then calculated by subtracting the accuracy at the baseline time point (e.g., baseline) from the accuracy at the later time points (e.g., immediately after treatment, 2 weeks post, and 2 months post). This reflects the change in the participant's ability to name trained items, expressed as absolute percent change. A positive difference indicates improvement in naming accuracy, with a larger change reflecting greater improvement. A negative difference indicates a decline, with a larger change reflecting greater deterioration in naming ability.
Time Frame: as for outcome 1
Population: Participants who completed oral naming.
Measure: Mean (Standard Deviation); unit: absolute percent change
Arm/Group | Active tDCS Plus Speech-Language Therapy | Sham Plus Speech-Language Therapy
Number analyzed (Participants) | 29 | 25
absolute percent change
  Phase 1: change from baseline immediately after treatment: number analyzed (Participants) | 14 | 15
  Phase 1: change from baseline immediately after treatment | 38.8 (7.3) | 26.9 (4.7)
  Phase 1: change from baseline 2-weeks post treatment: number analyzed (Participants) | 12 | 15
  Phase 1: change from baseline 2-weeks post treatment | 30 (7.5) | 21.3 (4.9)
  Phase 1: change from baseline 2-months post treatment. (Baseline for Phase 2): number analyzed (Participants) | 10 | 15
  Phase 1: change from baseline 2-months post treatment. (Baseline for Phase 2) | 24.9 (8.5) | 15.3 (4.8)
  Phase 2: change from baseline immediately after treatment: number analyzed (Participants) | 15 | 10
  Phase 2: change from baseline immediately after treatment | 23.5 (5.0) | 26.5 (10.9)
  Phase 2: change from baseline 2-weeks post treatment: number analyzed (Participants) | 15 | 9
  Phase 2: change from baseline 2-weeks post treatment | 15.6 (4.1) | 22.6 (8.9)
  Phase 2: change from baseline 2-months post treatment: number analyzed (Participants) | 14 | 10
  Phase 2: change from baseline 2-months post treatment | 6.5 (4.3) | 6.3 (6.3)

4. Primary Outcome: Absolute Percent Change in Oral Naming (Untrained Items)
Description: The percent accuracy for each participant's untrained oral naming list was calculated, with scores ranging from 0% to 100%. A score of 0% indicates no correct responses, while 100% represents perfect accuracy. Higher percentages reflect better performance. To assess changes in performance from pre- to post-treatment, the percent accuracy for untrained items was compared before and after the intervention. The absolute percentage change was then calculated by subtracting the accuracy at the baseline time point (e.g., baseline) from the accuracy at the later time points (e.g., immediately after treatment, 2 weeks post, and 2 months post). This reflects the change in the participant's ability to name trained items, expressed as absolute percent change. A positive difference indicates improvement in naming accuracy, with a larger change reflecting greater improvement. A negative difference indicates a decline, with a larger change reflecting greater deterioration in naming ability.
Time Frame: as for outcome 1
Population: Participants who completed oral naming.
Measure: Mean (Standard Deviation); unit: absolute percent change
Groups:
- Active HD-tDCS Plus Speech-Language Therapy: Active tDCS will be applied at the beginning of 45min speech-language therapy session and will last for 20 min.
  Active tDCS plus Speech-Language Therapy: Stimulation will be delivered by a battery-driven constant current stimulator. The electrical current will be administered to a pre-specified region of the brain (inferior frontal gyrus). The stimulation will be delivered at an intensity of 2mA (estimated current density 0.04 mA/cm2; estimated total charge 0.048C/cm2) in a ramp-like fashion for a maximum of 20 minutes. Speech-language therapy will be oral and written naming.
Arm/Group | Active HD-tDCS Plus Speech-Language Therapy | Sham Plus Speech-Language Therapy
Number analyzed (Participants) | 29 | 25
absolute percent change
  Phase 1: change from baseline immediately after treatment: number analyzed (Participants) | 14 | 15
  Phase 1: change from baseline immediately after treatment | 8.1 (2.4) | 8.9 (4.6)
  Phase 1: change from baseline 2-weeks post treatment: number analyzed (Participants) | 12 | 15
  Phase 1: change from baseline 2-weeks post treatment | 4.8 (2.5) | 7.9 (3.5)
  Phase 1: change from baseline 2-months post treatment. (Baseline for Phase 2): number analyzed (Participants) | 10 | 15
  Phase 1: change from baseline 2-months post treatment. (Baseline for Phase 2) | 3.9 (4.0) | 2.6 (4.6)
  Phase 2: change from baseline immediately after treatment: number analyzed (Participants) | 15 | 10
  Phase 2: change from baseline immediately after treatment | 4.8 (2.6) | -1.8 (7.2)
  Phase 2: change from baseline 2-weeks post treatment: number analyzed (Participants) | 15 | 9
  Phase 2: change from baseline 2-weeks post treatment | 1.8 (2.1) | 0.4 (2.9)
  Phase 2: change from baseline 2-months post treatment: number analyzed (Participants) | 14 | 10
  Phase 2: change from baseline 2-months post treatment | 4.6 (2.7) | -6.7 (3.8)

5. Secondary Outcome: Change in Sentence Comprehension as Measured by the Subject Object Active Passive (SOAP) Test
Description: The SOAP test is a test that has been shown to measure comprehension of simple and complex sentence structures. It contains sentences with different syntactic complexities: subject relatives, object relative, active and passive voice. The participant has to listen to a sentence and choose the correct picture that corresponds to its meaning amongst 3 alternatives. Scores range from 0-40 with higher scores indicating better comprehension. For each participant in each group absolute change from before to after treatment was calculated and the mean absolute change for the group was calculated.
Time Frame: Change from baseline to immediate follow-up (3 weeks).
Population: Participants who completed SOAP test
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active HD-tDCS Plus Speech-Language Therapy | Sham Plus Speech-Language Therapy
Number analyzed (Participants) | 12 | 17
score on a scale | 3.250 (3.911) | -0.412 (3.658)

6. Secondary Outcome: Change in Functional Connectivity
Description: Using resting-state functional magnetic resonance imaging (rsfMRI), investigators will investigate whether tDCS intervention will result in different changes in connectivity between the targeted area (left inferior frontal gyrus) and other nodes in the brain. Global connectivity is measured through the participation coefficient. The participation coefficient is scored on a scale from -1 to +1. Compared with healthy controls a score closer to +1 was associated with worse dementia severity.
Time Frame: Change from before treatment to immediate follow up (3 weeks)
Population: fMRI data were collected from 33 participants with PPA. One participant completed treatment but data was excluded due to rediagnosis. Analysis was only performed for period 1 of the intervention so only 16 participants with tDCS and 16 with sham are compared.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active HD-tDCS Plus Speech-Language Therapy | Sham Plus Speech-Language Therapy
Number analyzed (Participants) | 16 | 16
score on a scale | -0.08 (0.02) | 0.02 (0.01)
Statistical Analysis 1: Comparison: Active HD-tDCS Plus Speech-Language Therapy vs Sham Plus Speech-Language Therapy; Test type: Superiority; p < .05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were not assessed during the 12-week control condition (natural progression period) preceding treatment. Adverse events were assessed from randomization to up to 2 months post treatment for each intervention.
Arm/Group | Active HD-tDCS Plus Speech-Language Therapy | Sham Plus Speech-Language Therapy
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/32
Other Adverse Events (participants affected / at risk) | 0/36 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-08): https://cdn.clinicaltrials.gov/large-docs/22/NCT02606422/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-21): https://cdn.clinicaltrials.gov/large-docs/22/NCT02606422/ICF_001.pdf